CLINICAL TRIAL: NCT00569374
Title: Safety and Tolerability of Modafinil for Methamphetamine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Carole Hamon, University of Arkansas for Medical Sciences
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol / IRB # 79045
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Results first posted 2010-03-22 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-09

CONDITIONS: Methamphetamine Dependence
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Modafinil — subjects attend clinic for the first week in order to receive meds; oral, 200mg/day doses for three days for initiation doses; increased to oral 400mg/day for the remainder of the trial (weeks 2-6); washout period during week 7

SUMMARY:
This 7 week, open-label pilot clinical trial will examine the safety and tolerability of modafinil up to 400mg/day as a potential treatment to reduce methamphetamine use in methamphetamine-dependent volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* not currently enrolled in a treatment program
* subjects must have a history of methamphetamine use with recent use confirmed by a positive urine toxicology screen for amphetamines during the month prior to study entry
* subjects must meet DSM-IV criteria for amphetamine dependence as assessed by the substance abuse section of the Structured Clinical Interview for DSM-IV (SCID)
* women of childbearing age must have a negative pregnancy test to enroll in this study, agree to monthly pregnancy testing, and agree to use appropriate forms of birth control for the duration of the study

Exclusion Criteria:

* current diagnosis of alcohol, opiate, or sedative physical dependence
* ill health (e.g., major cardiovascular, renal, endocrine, hepatic disorder)
* history of schizophrenia, or bipolar type I disorder
* present or recent use of over-the-counter or prescription psychoactive drug or drug(s) that would be expected to have major interaction with drug to be tested
* medical contraindication to receiving study medications (e.g., allergy to modafinil, treatment with cyclosporine, clomipramine, or desipramine)
* Current suicidality or psychosis
* liver function tests (i.e., liver enzymes) greater than three times normal levels
* pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Janette McGaugh, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Modafinil: All participants were started on Modafinil titrated to 400mg in this open label trial.
Period: Overall Study
Arm/Group | Modafinil
Started | 8
Completed | 4
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Modafinil
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 45.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: Heart rate as a safety measure was measured by thrice weekly measuring heart rate in beats per minute.
Time Frame: Thrice weekly for 7 weeks
Population: The data reported was obtained by computing the overall mean heart rate for each participant, then using these to compute the overall mean.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Modafinil
Number analyzed (Participants) | 8
beats per minute | 79.66 (2.22)

2. Primary Outcome: Systolic Blood Pressure
Description: Systolic blood pressure as a safety measure was measured by thrice weekly measuring blood pressure in mmHg.
Time Frame: Thrice weekly for 7 weeks
Population: The data reported was obtained by computing the overall mean systolic blood pressure for each participant, then using these to compute the overall mean.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Modafinil
Number analyzed (Participants) | 8
mmHg | 128.62 (3.15)

3. Primary Outcome: Diastolic Blood Pressure
Description: Diastolic blood pressure as a safety measure was measured by thrice weekly measuring blood pressure in mmHg.
Time Frame: Thrice weekly for 7 weeks
Population: The data reported was obtained by computing the overall mean diastolic blood pressure for each participant, then using these to compute the overall mean.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Modafinil
Number analyzed (Participants) | 8
mmHg | 81.49 (2.67)

4. Primary Outcome: "Modafinil Side Effects Checklist"
Description: Modafinil side effects were measured weekly by means of the Modafinil Side Effects Checklist which asked participants to rate their experience of the following potential side effects: headaches, nausea, nervousness, runny nose, diarrhea, back pain, anxiety, insomnia, dizziness and upset stomach. Participants rated their experience on a 4 point scale ranging from "not at all" (0) to "very much (4). The score was determined by units on a scale.
Time Frame: Weekly for 7 weeks
Population: The data reported was obtainined by computing the overall mean numberical score on the Modafinil Side Effects Checklist for each participant, then using these to compute the overall mean. The checklist is a 10 item scale with each item scoring between 0 (none) to 4 (worst). The potential scores range from 0 (least) to 40 (worst).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil
Number analyzed (Participants) | 8
units on a scale | 3.75 (2.94)

5. Primary Outcome: Anxiety as Measured by the Hamilton Anxiety Scale
Description: Participants were administered the Hamilton Anxiety Scale thrice weekly throughout the study. The scale is a 14 item questionaire with scores ranging from 0 to 56.
Time Frame: Thrice weekly for 7 weeks
Population: The data reported was obtained by computing the overall mean score on the Hamilton Anxiety Scale for each participant, then using these to compute the overall mean. The scale is a 14 item instrument with each item scoring a potential range of 0 (none) to 4 (worst). The potential total scores range form 0 (least) to 56 (worst).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil
Number analyzed (Participants) | 8
units on a scale | 4.07 (2.44)

6. Primary Outcome: Depression as Measured by the Hamilton Depression Scale
Description: Participants were administered the Hamilton Depression Scale thrice weekly throughout the study. The scale is a 21 item questionaire with scores ranging from 0 to 62 with a cutoff for depression of 15.
Time Frame: Thrice weekly for 7 weeks
Population: The data reported was obtained by computing the overall mean score on the Hamilton Depression Scale for each participant, then using these to compute the overall mean. It is a 22 item scale of which 13 items have a score of 0 (none) to 4 (worst) and 9 have a score of 0 (none) to 2 (worst). The total score ranges from 0 (least) to 70 (worst).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil
Number analyzed (Participants) | 8
units on a scale | 5.64 (3.41)

7. Secondary Outcome: Methamphetamine Withdrawal as Measured Using the Amphetamine Withdrawal Questionaire.
Description: The Amphetamine Withdrawal Questionaire was given at intake and 3 times weekly during the first 3 weeks of the study. This time span was chosen due to the tendency of methamphetamine withdrawal to enter an acute phase in the first week after last use with a subsequent subacute phase following for the next two weeks(McGregor et al, 2005). This questionaire is comprised of 10 items which describe symptoms associated with the cessation of chronic amphetamine use for which participants indicate severity on a 4-point scale. The minimum score is 0 and the maximum score is 40.
Time Frame: Thrice weekly for the first three weeks
Population: The data reported was obtained by computing the overall mean numerical score on the Amphetamine Withdrawal Questionaire for each participant, then using these to compute the overall mean. The scale consists of 13 items ranging from 0 (none) to 4 (worst). The total score ranges from 0 (least) to 52 (worst).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Modafinil
Number analyzed (Participants) | 8
units on a scale | 5.79 (4.42)

ADVERSE EVENTS:
Time Frame: These results were collected over a period of 1 year and 10 months. Five Adverse events occurred during the study, of which three were probably related to study participation.
Description: Adverse events included one report each of tachycardia and dry mouth. The third occurred when a subject missed a dose on one day and took a double dose the next day. The subject experienced tachycardia, dry mouth, nervousness which resolved within one hour of modafinil ingestion.
Arm/Group | Modafinil
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modafinil (N=8)
Tachycardia (General disorders) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Tachycardia, dry mouth, nervousness after taking extra dose (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes